CLINICAL TRIAL: NCT05796258
Title: A Multi-institutional Effort With a Three-pronged Centralized Molecular Analysis to Optimize Detection of NTRK1,2,3 Fusions in Thyroid Cancer
Brief Title: Three-pronged Centralized Molecular Analysis to Optimize Detection of NTRK1,2,3 Fusions in Thyroid Cancer
Acronym: NTRK
Status: Completed | Type: Observational
Sponsor: Regina Elena Cancer Institute (Other)
Collaborators: University of Roma La Sapienza (Other); Bambino Gesù Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Marialuisa Appetecchia, Professor, Regina Elena Cancer Institute
Other Study IDs: RS1445/20(2421)
Record Dates: First submitted 2023-03-16; First posted 2023-04-03 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Thyroid Cancer
Keywords: ntrk fusion
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor tissue is routinely obtained after the surgical removal of the tumor tissue (primary or metastatic).
  Part of the tissue will be immediately processed for RNA extraction, the rest of the tissue is processed for conventional histology/IHC analysis and stored in the institutional tissue biobank.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: NTRK fusion assessment — To evaluate NTRK fusion presence by MCG, Immunohistochemistry or NGS

SUMMARY:
This multi-center study aims at NTRK fusion testing of all patients with advanced thyroid cancer (any histotype and regardless of stage). The primary objective of this study is to assess the frequency of NTRK fusions in thyroid cancer. The secondary objective of this study is to develop an effective tool (testing) strategy for the detection of NTRK fusions in thyroid tumors, comparing the diagnostic tecniques available (IHC, real-time PCR and NGS).

DETAILED DESCRIPTION:
Thyroid cancer is the most common neoplasm of the endocrine system. Most thyroid carcinomas originate from the follicular epithelium and are distinguished in differentiated forms (DTC): papillary (PTC) and follicular (FTC) carcinomas. Both have a favorable prognosis and account for approximately 80% and 10% of all thyroid neoplasms, respectively. The undifferentiated form represented by the anaplastic thyroid carcinoma (ATC) is less frequent (about 2%) and represents one of the most aggressive human tumors with a survival that rarely exceeds 6-12 months. Medullary thyroid carcinoma (MTC), deriving from parafollicular C cells, is relatively rare (approximately 5%) and is associated with an intermediate prognosis between differentiated and poorly differentiated forms.

As to the prevalence of NTRK lesions, many authoritative papers and reviews claim very high (up to 75%) NTRK fusion frequencies, particularly in the common PTC. However, an extensive PubMed analysis back to year 1990 does not provide convincing support for this claim.Several techniques for NTRK fusion diagnosis exist, including pan-Trk IHC, FISH, reverse transcription PCR, DNA-based next-generation sequencing (NGS), and RNA-based NGS. Each of these assays has unique features, advantages, and limitations, and familiarity with these assays is critical to appropriately screen for NTRK fusions.

The aim of this study is to determine the frequency of NTRK fusions in advanced thyroid cancer patients and to compare the diagnostic tecniques available (IHC, real-time PCR and NGS).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced thyroid cancer (any histotype)
* Informed consent.

Exclusion Criteria:

* Patients with thyroid neoplasms without appropriate material for subsequent immunohistochemical and molecular studies;
* Patients with non-advanced thyroid cancer

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients affected by advanced thyroid cancer (any histotype)
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-04 (Actual)

PRIMARY OUTCOMES:
Frequency of NTRK fusions in thyroid cancer | from 01-Jan-2022 to 31-Dec-2023
  To assess the frequency of NTRK fusions in histological sample of tumors by patients affected by thyroid cancer, assessed as the number of tumor harboring NTRK fusion on the total of tumor analized

SECONDARY OUTCOMES:
Assesment of the ability of Immunohistochemistry to identify for NTRK fusion | from 01-Jan-2022 to 31-Dec-2023
  To assess the ability of Immunohistochemistry to detect NTRK fusion on histological sample (using NGS as comparator)
Assesment of the ability of real time PCR to identify for NTRK fusion | from 01-Jan-2022 to 31-Dec-2023
  To assess the ability of real time PCR to detect NTRK fusion on histological sample (using NGS as comparator)

CONTACTS AND LOCATIONS:
Overall Officials: Marialuisa Appetecchia, Prof, Principal Investigator — Regina Elena Cancer Institute
Locations (1):
- Regina Elena National Cancer Institute, Roma, Italy

IPD SHARING:
Plan to Share IPD: Yes
Raw data will be published in open access databases
Supporting Information: Study Protocol, Analytic Code
Time Frame: After study end
Access Criteria: open access
URL: http://garr.it